CLINICAL TRIAL: NCT06684964
Title: Real-World Evidence Non-interventional Prospective Study for the Effectiveness, Tolerability and Adherence of Asciminib After Two Previous TKIs in Patients With Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) in Saudi Arabia. (ASC4REAL)
Brief Title: RWE,NIS,Prospective Study for the Effectiveness, Tolerability and Adherence of Asciminib in Saudi Arabia. (ASC4REAL)
Acronym: ASC4REAL
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001ASA01
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Chronic Myelogenous Leukemia in Chronic Phase
Keywords: Chronic Myelogenous Leukemia in chronic phase; CML-CP; Asciminib
MeSH Terms: interventions — asciminib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Asciminib: Patients who have been receiving asciminib for up to 6 months prior to study start
  Interventions: Other: asciminib

INTERVENTIONS:
Other: asciminib — This is an observational study. There is no treatment allocation. The decision to initiate asciminib will be based solely on clinical judgement.

SUMMARY:
This is a non-interventional, prospective, observational single arm study describing the real-world effectiveness, tolerability, adherence, Healthcare Resource Utilization (HCRU) and Patient-Reported Outcome (PRO) data of asciminib in patients with Ph+ Chronic Myelogenous Leukemia - Chronic Phase (CML-CP) previously treated with ≥2 Tyrosine Kinase Inhibitor (TKIs) in routine clinical practice in Kingdom of Saudi Arabia.

DETAILED DESCRIPTION:
Patients who have been receiving asciminib for up to 6 months prior to study start will be enrolled over a period of approximately 6 months and followed up for 12 months to assess study outcomes.

Each patient will be followed from baseline up to the earliest of death, loss to follow-up or end of the 12-month follow-up.

The study aims to enrol approximately 40 patients in a single arm design from a total of 6 centers in Kingdom of Saudi Arabia (KSA) over an enrollment period of approximately 6 months. These patients must have been prescribed asciminib for a maximum of 6 months before enrolling in the study. The prescription of asciminib should align with its approved label use. Importantly, the decision to prescribe asciminib to these patients should have been made independently by the physician and not influenced by the study. Data will be collected from patient electronic medical records in the sites chosen.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet all the following criteria:

1. Signed and dated Patient Informed Consent Form obtained.
2. Male or female patients with a diagnosis of Ph+ CML-CP ≥18 years of age with the following laboratory values:

   1. <15% blasts in peripheral blood and bone marrow
   2. <30% blasts plus promyelocytes in peripheral blood and bone marrow
   3. <20% basophils in the peripheral blood
   4. ≥50 x 109/L (≥50,000/mm3) platelets

4. Prior treatment with a minimum of 2 prior TKIs: e. First-generation TKI imatinib f. 2G-TKI dasatinib, nilotinib and bosutinib g. 3G-TKI ponatinib 4. Patients are currently receiving asciminib as per approved local label and independently of study participation. Patients must have started asciminib therapy no more than 6 months prior to their enrollment in the study.

Exclusion Criteria:

Patients meeting ANY of the following criteria are not eligible for participation:

1. Asciminib based treatment regimen in first or second line.
2. Patients are currently participating in any other clinical trials.
3. Patients who refused to sign informed consent.
4. According to the investigator's opinion, the patient is an unlikely candidate to provide an accurate medical history and/or to obtain long-term follow-up information for any reasons such as unavailability or severe concomitant illnesses.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have been prescribed asciminib for a maximum of 6 months before enrolling in the study. Patients will be included in the study regardless of their MMR status at the initiation of asciminib treatment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Major molecular response (MMR) | Month 12
  MMR is defined as a breakpoint cluster region-Abelson murine leukemia viral oncogene homolog 1 protein (BCR-ABL1) transcript level ≤0.1%, at 12 months.

SECONDARY OUTCOMES:
Frequency and severity of hematologic and non-hematologic AEs | Up to 12 months
  Frequency and severity of hematologic and non-hematologic AEs
Major Molecular Response (MMR) Rate | Baseline, month 6, month 12
  MMR is defined as a BCR-ABL1 transcript level ≤0.1%.
Deep Molecular Response (DMR) Rate | Month 6, month 12
  Percentage of participants with MR4.0 and MR4.5:
  * MR4.0 [ BCR-ABL1 transcript level ≤0.01%]
  * MR4.5 [ BCR-ABL1 transcript level ≤0.0032%]
Cytogenetic Response (CCyR) Rate | Month 6, month 12
  Assessment of CCyR and/or [BCR-ABL1 transcript level ≤1%]
Duration of MMR | Up to 12 months
  Assess the duration of MMR in participants.
Simplified Medication Adherence Questionnaire (SMAQ) score. | Month 6, month 12
  SMAQ assesses adherence to medication. It is a 6-item questionnaire that evaluates different aspects of patient compliance with treatment: forgetfulness, routine, adverse effects, and omissions. A patient is classified as non-compliant if he/she responds to any of the questions with a non-adherence answer, and in terms of quantification, if the patient has lost more than two doses during the last week or has not taken medication during more than two complete days during the last three months.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Saudi Arabia (3):
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh

IPD SHARING:
Plan to Share IPD: No